CLINICAL TRIAL: NCT06436118
Title: Evaluation of the Use of the RELAX® Glasses on the Anxiety of Patients Undergoing Emergency Hand Surgery Under Locoregional Anesthesia Compared to Those Who do Not Use the Glasses
Brief Title: Evaluation of the Use of the RELAX® Glasses on the Anxiety of Patients Undergoing Emergency Hand Surgery Under Locoregional Anesthesia
Acronym: RELAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Valenciennes (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-05
Record Dates: First submitted 2022-08-29; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Surgery
Keywords: Audiovisual sedation; anxiety; hand surgery; locoregional anesthesia
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with RELAX® glasses (Experimental)
  Interventions: Behavioral: RELAX® glasses
- Group without RELAX® glasses (No Intervention)

INTERVENTIONS:
Behavioral: RELAX® glasses — Glasses which are a solution of audiovisual sedation by positive distraction for hospital medical use.
  Arms: Group with RELAX® glasses

SUMMARY:
More than 90% of hand surgery is performed under local anesthesia and can be a source of anxiety, especially in an emergency context. The management of this intraoperative anxiety is essential for the comfort. The use of a virtual reality headset has shown its effectiveness in reducing anxiety in dental surgery or hand surgery under local anesthesia with the WALANT technique. On the other hand, virtual reality and the use of 3D can cause discomfort and side effects such as nausea and dizziness. It is known that audiovisual distraction also effectively reduces pain and anxiety in patients with fewer side effects.

The investigators have therefore chosen to use the RELAX® glasses. There are no publications examining the effectiveness of positive distraction as a non-pharmacological agent to improve the patient experience during emergency management in the operating room in the context of hand surgery under locoregional anesthesia. The investigatos would like to study its action on the anxiety, pain and global satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for hand surgery under emergency locoregional anesthesia (Wounds, fractures and infections of the hand and wrist).
* Over 15 years and 3 months of age on the day of inclusion.
* Patient with written consent or additional parental consent in the case of minor patients.
* Socially insured patient.
* Patient willing to comply with all study procedures and duration.

Exclusion Criteria:

* Medical history contraindicating RELAX glasses: claustrophobia.
* Known and current alcohol and/or illicit drug abuse that may interfere with patient safety and/or compliance.
* Any condition that would make the patient unfit for the study: current presence of cognitive impairment (MMS <15), severe psychiatric disorders (bipolar disorder, psychotic disorders according to the DSM-V classification).
* Pregnant or breastfeeding woman.
* Patient under court protection.
* Patient participating in another study.
* Patient's refusal to use the headset.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in visual analogue scale anxiety scores after emergency hand surgery | In the 5 minutes after the end of emergency hand surgery
  The visual analogue anxiety scale from 0 to 10, with 0 meaning no anxiety and 10 very high anxiety.

SECONDARY OUTCOMES:
Overall satisfaction between the group using RELAX glasses and the group following the usual course (without RELAX glasses) measured by a visual analogue scale | Immediate postoperative
  The visual analogue satisfaction scale ranges from 0 to 10, with 0 meaning unsatisfaction and 10 indicating very high satisfaction.
Variation in pain between entering and leaving the operating theatre between the 2 arms using a visual analogue scale | In the 5 minutes after the end of emergency hand surgery
  The visual analogue pain scale ranges from 0 to 10, with 0 meaning non pain and 10 meaning very high pain
Rate of patients receiving at least one additional analgesic | Immediate after locoregional anaesthesia
Rate of patients receiving at least one additional anxiolytic | Immediate after locoregional anaesthesia
Pre-existing anxiety, only in patients receiving RELAX glasses, measured with the STAI-YB score | 7-days after emergency hand surgery
  Only in patients receiving RELAX glasses : If the STAI-YB score is higher than 65, the patient is considered to have pre-existing anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Valenciennes, Valenciennes, France